CLINICAL TRIAL: NCT04121546
Title: Collaborative Care for Opioid Dependence And Pain Pilot Study
Acronym: CCODAPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Indiana University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Michael A. Bushey, Assistant Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1905213338; KL2TR002530 (NIH)
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Results first posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Opioid Dependence; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients will receive the telecare intervention.
  Interventions: Behavioral: Telecare Intervention
- Usual Care Arm (No Intervention): Patients will receive usual care.

INTERVENTIONS:
Behavioral: Telecare Intervention — Patients will meet with a care coordinator to discuss current opioid use pattern and potential reduction strategies. Participants will fill out baseline measures. A 6 week positive psychology intervention will also be introduced in which patients will practice different techniques each week over 6 weeks, and will then practice incorporating a single technique into daily practice for the remaining 6 weeks. During the first 6 weeks, patients will have weekly check in meetings with a care manager to report on any withdrawal symptoms. These meetings will space to ever other week during the remaining 6 weeks. Possible treatment adjustments will be discussed between the care coordinator and primary investigator at weekly meetings. At the completion of the 12 week study, patients will complete outcome measures.
  Arms: Intervention Arm

SUMMARY:
This pilot study evaluates a collaborative care program to assist with opioid tapering in patients with chronic pain. Patients will be randomized to receive the intervention or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain for at least 6 months
* Receiving daily opioid treatment

Exclusion Criteria:

* Not speaking English
* Significant psychiatric impairment including severe cognitive impairment, suicidality, schizophrenia, or bipolar disorder
* Known life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Bushey, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Usual Care Arm
Started | 2 | 4
Completed | 1 | 1
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 2 | 4 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (12.7) | 61.0 (6.8) | 57.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 4 | 6
Opioid Dose [Mean (Standard Deviation); unit: Morphine Milligram Equivalents] | 35.0 (35.4) | 27.5 (21.8) | 30 (23.5)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Dose Change
Description: Percentage change in daily opioid morphine milligram equivalent (MME) dose
Time Frame: 12 weeks
Population: Participants who completed the 12 week survey were included for analysis.
Measure: Mean (Full Range); unit: percentage of MME reduction
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 1 | 1
percentage of MME reduction | 62.5 [62.5 to 62.5] | 50 [50 to 50]

2. Secondary Outcome: Change in PROMIS Pain Interference
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.1 - Pain Interference 8a is an 8-item scale from the PROMIS item bank which assesses self-reported consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Each item has a 5-point Likert response, with total scores ranging from 8 - 40, with higher numbers corresponding to worse pain interference outcomes. For this outcome, the score at baseline was subtracted from the score at 12 weeks to determine the change score, with negative change scores demonstrating symptom improvement (i.e. less pain interference).
Time Frame: 12 weeks
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 1 | 1
scores on a scale | -0.25 [-0.25 to -0.25] | -0.63 [-0.63 to -0.63]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intervention Arm | Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4
Other Adverse Events (participants affected / at risk) | 1/2 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=2) | Usual Care Arm (N=4)
opioid withdrawal (Psychiatric disorders) | 1 (1) | 0 (0) — Participant experienced mild symptoms of opioid withdrawal

LIMITATIONS AND CAVEATS:
Due to the low rate of enrollment/completion, the design was determined to be infeasible and the trial was ended early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT04121546/Prot_SAP_000.pdf